CLINICAL TRIAL: NCT03251352
Title: Tyrosine Kinase Inhibitor Discontinuation in Adults Patients With Chronic Myeloid Leukemia in China
Brief Title: TKI Discontinuation in CML Patients of China
Acronym: TFR_china
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201733572018022
Record Dates: First submitted 2017-05-07; First posted 2017-08-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-06

CONDITIONS: Leukemia; Myelogenous; Chronic; BCR-ABL (Breakpoint Cluster Region-abelson Murine Leukemia); Positive
Keywords: TKI, CML, discontinuation
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TKI Discontinuation Group: The enrolled patients will be undertaking TKI discontinuation under the conditions of informed consent and frequent monitoring according to the clinical guideline.

SUMMARY:
The primary objective of this study is to describe the maintenance of the molecular remission after tyrosine kinase inhibitor (TKI) disconnection in chronic myeloid leukaemia (CML) patients in China in the real-world clinical practice setting. This is a post-marketing, non-interventional, single-arm, prospective registry study in adult patients with chronic phase (CP) and accelerated phase (AP) in China. Patients will be recruited consecutively from the study sites during the enrollment period. The enrolled patients will be undertaking TKI discontinuation under the conditions of informed consent and frequent monitoring according to the clinical guideline.

DETAILED DESCRIPTION:
Tyrosine kinase inhibitors (TKIs) are the standard of care for patients with chronic myeloid leukaemia (CML) in chronic phase. Imatinib, the first ATP competitive TKI, received approval for use based on a dramatic and durable survival benefit. Other TKIs, the second generation compounds dasatinib, nilotinib and bosutinib and the third generation drug ponatinib, were designed and tested for a greater target-specific potency. With the development of these effective TKI treatments, CML disease burden can be reduced to minimal levels, and CML patients can have a life expectancy similar to that of the general population. Although TKI treatment may result in a deep, stable molecular remission, CML treatment guidelines recommend that patients continue TKI treatment indefinitely. However, Chronic TKI therapy can cause drug-related adverse reactions and constitute financial difficulties, which can result in decreased adherence to therapy. Therefore, the concept of a lifelong therapy with TKIs has thus been challenged and treatment-free remission (TFR) strategies will soon integrate clinical practice.TFR can be defined as the ability to maintain molecular remission without taking any TKI therapy. Studies have demonstrated the feasibility of successful TFR. In the STIM and TWISTER trials, imatinib discontinuation was proposed providing that patients had achieved deep molecular response for a certain period. The 2-year probability to maintain such deep molecular response levels without any TKI therapy was 38% in STIM and 47% in TWISTER. Subsequently, several studies were conducted and confirmed that imatinib-free remission was possible. Discontinuation of new generation TKIs was also investigated and indicated that dasatinib or nilotinib may promote access to TFR strategies as compared to imatinib. TFR is on the way to become an important goal in clinical practice, implicating an alternation in CML management guidelines in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Adults with CML-CP/AP and willingness of TKI discontinuation;
* With ≥ 5 years frontline imatinib, reached MMR (major molecular response) in 2 years, with ≥ 2 years MR (molecular response) 4.5;
* Reached MMR with frontline imatinib, with ≥ 2 years nilotinib, with ≥ 1 year MR4.5;
* Failure with frontline imatinib, reached MMR in 1 year with nilotinib, with ≥ 2 years MR4.5;
* With ≥ 3 years frontline imatinib, reached MMR in 1 year, with ≥ 2 years MR4.5.

Exclusion Criteria:

* Diagnosed with CML-BP before TKI treatment;
* With a TKI discontinuation of over 30 days in the first year;
* With a TKI discontinuation of over 30days on average annually;
* Reduced the dosage of TKI treatment without instructions;
* Transferred to the second-generation TKIs after resistance to imatinib.
* Under the treatment of stem cells transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population is CML patients under TKI treatment in China.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Molecular Remission Rate | at 12 months
  The molecular remission rate

SECONDARY OUTCOMES:
Adverse Events | through study completion, an average of 1 year
  Incidence of Treatment-free related Adverse Events
Recurrence | through study completion, an average of 1 year
  CML molecular recurrence
QoL | through study completion, an average of 1 year
  EROTC-QLQ-C30 and EROTC-QLQ-CML-24

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No